CLINICAL TRIAL: NCT01993654
Title: In Vivo Confocal Microscopy Study of Pigmented Conjunctival Lesions
Status: Terminated | Type: Observational
Why Stopped: Study was terminated due to low recruitment.
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Wills Eye (Other)
Responsible Party: Sponsor
Other Study IDs: 09-04-028
Record Dates: First submitted 2011-10-19; First posted 2013-11-25 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Nevus; Racial Melanosis; Primary Acquired Melanosis; Conjunctival Malignant Melanoma
Keywords: Pigmented Lesions; PAM; Ocular lesion
MeSH Terms: conditions — Nevus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Nevus
  Interventions: Procedure: HRT III with Non-Contact Cornea Rostock Module
- Racial Melanosis
  Interventions: Procedure: HRT III with Non-Contact Cornea Rostock Module
- Primary Acquired Melanosis
  Interventions: Procedure: HRT III with Non-Contact Cornea Rostock Module
- Malignant Melanoma
  Interventions: Procedure: HRT III with Non-Contact Cornea Rostock Module
- Normal
  Interventions: Procedure: HRT III with Non-Contact Cornea Rostock Module

INTERVENTIONS:
Procedure: HRT III with Non-Contact Cornea Rostock Module — Confocal imaging of the conjunctival lesion

SUMMARY:
This study aims to validate the use of laser in vivo confocal microscopy as an early diagnostic and differentiation tool of pigmented conjunctival lesions, evaluate the efficacy of in vivo confocal microscopy for follow-up (as a visualizing tool) after tumor resection for early detection of tumor recurrence, and to evaluate the use of in vivo confocal microscopy in evaluation of response to treatment. The modified technique with Heidelberg Retina Tomography (HRT) confocal microscopy and anterior segment optical coherence tomography (OCT) are non-invasive, no-touch, imaging techniques that may help in differentiation of benign lesions like nevi or racial melanosis, from malignant lesions like primary acquired melanosis and malignant melanomas. The OCT will potentially allow to estimate tumor depth in vivo as preliminary studies have shown.

DETAILED DESCRIPTION:
Conjunctival melanoma is a potentially lethal neoplasm, with an average 10-year mortality rate of 30%, and 15-year mortality rate of 45%. This condition occurs mainly in the white population, with rare reports in black and other non-white populations. Recent studies have indicated that like cutaneous melanoma, the incidence of conjunctival melanoma is increasing.

Conjunctival Malignant Melanoma (MM) is also currently diagnosed based upon clinical grounds, through observation of the growth of the suspected lesions over regular intervals of time. Unfortunately simple slit lamp examination is currently the only clinical diagnostic visual instrument available in medical practice, and the early diagnosis of MM by slit-lamp examination is still rather poor. Further the diagnosis of invasive conjunctival MM is currently established by conjunctival excisional biopsy and defined by the invasion of the underlying substantia propria of the conjunctiva by atypical tumor cells, especially when there is loss of the maturation. Regarding the management of malignant melanoma, unfortunately the extensive horizontal and even vertical growth of this neoplasm does not always lend itself to simple excision leading to exenteration. As a vision-sparing alternative, local excision with cryotherapy has become the treatment of choice. Long-term follow-up has shown that local recurrences are common. More recently, topical chemotherapy with mitomycin C (MMC) has been used to treat cases with extensive PAM with atypia , because the pigmented margin is used as a guide for most conservative treatments, the tumor's edge may be missed.

Recurrent conjunctival MM often presents as an amelanotic mass and may be mistaken for pyogenic granuloma in a patient who has had multiple previous excisions of conjunctival MM, even though the original tumor may have been pigmented. Because of the lack of pigment, these tumors can remain unrecognized and progressively enlarge, especially if the patient has had previous surgery and conjunctival scarring. In addition, the tumor margins of recurrent amelanotic conjunctival MM may be indistinct. These factors can lead to delayed recognition and the unnecessary need for exenteration. Despite these radical procedures, which usually lead to loss of vision or the eye, these patients have been shown to have a poor survival rate, suggesting that metastasis has already occurred at the time of treatment. This confirms that the extent of the disease at diagnosis is the most important factor to determine the outcome. Recurrence of conjunctival MM is reported at 26% at 5 years and, 51% at 10 years.

MM of the conjunctival represents one of the greatest challenges in early or preventive detection. Whereas surgical excision in early stages of tumor development is almost always curative, delayed recognition puts the patient at risk of destructive growth and death once the tumor has progressed to competence for metastasis. Accurate diagnosis of pigmented lesions of the conjunctiva such as nevi, primary, and secondary acquired melanosis and MM present a challenge to both the ophthalmologist and the pathologist. It is not possible clinically to distinguish between PAM with and without atypia. The ability to detect early MM remains of paramount importance in our efforts to curtail deaths related to this malignancy. The implementation and utilization of in vivo imaging technologies in clinical practice would enhance our ability to detect MM while this cancer is in its early stages and curable. Further, accurate assessment of therapeutic tumor response is critical for evaluation of chemotherapy results in patients, and in clinical trials. Tumor response is also a guide for the clinician and patient or study. Early, accurate prediction of non-response would allow an early change to second-line treatment, thus sparing patient's unnecessary toxicity, psychological morbidity and delay of initiation of effective treatment. These are very few variables that investigators, as clinicians, can control regarding the management of conjunctival MM. However, early detection, technique and time of surgery may ultimate after tumor recurrence, need for orbital exenteration, tumor metastasis, and patient death. This non-invasive imaging technique that is now available for clinical studies might help in early detecting and preventing above mentioned problems.

ELIGIBILITY:
Inclusion criteria:

1. Age over 18 years
2. The ability to provide informed consent for enrollment in the study
3. Diagnosis of conjunctival nevus (Group 1 only)
4. Diagnosis of racial melanosis (Group 2 only)
5. Diagnosis or suspicion of primary acquired melanosis (PAM), scheduled for biopsy (Group 3 only)
6. Diagnosis of possible MM scheduled for biopsy (Group 4 only)
7. Confirmed diagnosis of MM based upon clinical and histopathological findings, and have already undergone resection(Group 4 only)
8. Confirmed diagnosis of MM recurrence based upon clinical and histopathological findings(Group 4 only)
9. Clear cornea (Group 5 only)
10. No conjunctival lesions or recent conjunctival diseases(Group 5 only)
11. No recent chemotherapy or radiotherapy(Group 5 only)

Exclusion criteria:

1. History of previous ocular surgery within last 3 months
2. History of inflammatory eye diseases within last 3 months
3. Current or history of glaucoma disease and on glaucoma medication
4. Contact lens use within last 3 months
5. Physical inability to cooperate for confocal microscopy
6. Prior history of infectious keratitis within 3 months
7. Suspicion for PAM or malignant melanoma (MM)(Groups 1,2,3)
8. History of PAM or MM(Groups 1,2,3)
9. Histopathology not confirmatory for MM (group 4 only)
10. History of other ocular carcinoma or any recent ocular topical chemotherapy or radiotherapy (Group 5 only)
11. History of cancer elsewhere in the body which is currently under systemic chemotherapy (group 5 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients over the age of 18 and belonging to one of the following groups will be recruited for this study.
  Group 1: Nevus Group 2: Racial melanosis Group 3: Primary Acquired Melanosis Group 4: Malignant Melanoma of the Conjunctiva Group 5: Normal Subjects with no pigmented lesions Normal subjects will be recruited from patients normally seen during clinic for cataract evaluations. Groups 1-4 will be identified by the investigators at MEEI and other 2 sites as potential study subjects during regular clinic visits.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Pigmented conjunctival lesions | Day 1
  Heidelberg Retina Tomography (HRT) and Optical Coherence Tomography (OCT) will be used to measure pigmented conjunctival lesions. (HRT) is performed with a confocal scanning laser ophthalmoscope. Along with corneal analysis software, the HRT is able to image cells and cell layers within the cornea. Optical Coherence Tomography (OCT) is a noninvasive optical imaging modality analogous to an ultrasound B-scan. OCT images will be used to estimate tumor depth.
  Immunohistochemistry results will be recorded from stained tissue samples obtained during surgical resections scheduled for study subjects with newly diagnosed conjunctival lesions. These patients will have HRT and OCT imaging performed prior to their standard of care surgery to remove the conjunctival lesion. Histologic and immunohistochemistry results and clinicopathologic findings will be analyzed by two observers and correlated with IVCM and OCT images of the same lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Hamrah, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary; Carol Shields, MD, Principal Investigator — Wills Eye Hospital; Arman Mashayekhi, MD, Principal Investigator — Wills Eye Hospital; Bita Esmaeli, MA, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Massachusetts Eye & Ear Infirmary, Boston, Massachusetts
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Study data was not analyzed due to sample size and no statistical power.